CLINICAL TRIAL: NCT05514769
Title: Proximal Gastrectomy Anterior Anastomosis With Pyloroplasty Versus Esophagogastric Anastomosis for Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Yunhong Tian, Professor, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220720
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Proximal Gastric Adenocarcinoma; Gastric Cancer; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Stomach Neoplasms; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal Gastrectomy Anterior Anastomosis With Pyloroplasty (GAP) (Experimental): The reconstruction including esophagogastric anastomosis and pyloroplasty for patients who underwent proximal gastrectomy . The anastomosis locate in the anterior of gastric stump.
  Interventions: Procedure: Proximal Gastrectomy Anterior Anastomosis With Pyloroplasty
- Control (Active Comparator): The reconstruction including esophagogastric anastomosis and pyloroplasty for patients who underwent proximal gastrectomy . The anastomosis locate in the posterior or side of gastric stump.
  Interventions: Procedure: Proximal Gastrectomy Anterior Anastomosis With Pyloroplasty

INTERVENTIONS:
Procedure: Proximal Gastrectomy Anterior Anastomosis With Pyloroplasty — The location of the anastomosis in the anterior of the gastric stump. Pyloroplasty is added in the procedure

SUMMARY:
This research is designed to compare proximal gastrectomy anterior anastomosis with pyloroplasty with esophagogastric anastomosis for gastric cancer. Gastroesophageal reflux disease, postoperative quality of life, short term outcomes, and long term outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the stomach, T1-T4 stages.
2. Eastern Cooperative Oncology Group performance status of 0 or 1.
3. Adequate organ function.

Exclusion Criteria:

1. Patients had distant metastasis.
2. oesophageal invasion of more than 3 cm.
3. Borrmann type 4 or large (more than 8 cm) type 3 carcinoma.
4. Previous chemotherapy or radiation therapy for any other malignancies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastroesophagus reflux disease apprised by ph monitoring | 6 months
  Ph monitoring by wireless or wire device
Gastroesophagus reflux disease apprised by questionnaire | 6 months
  PGSAS-45 questionnaire is adopted.

SECONDARY OUTCOMES:
Surgical complications of proximal gastrectomy for gastric cancer | 1 year
  Surgical complications include anastomotic leakage, anastomotic stricture, postoperative bleeding, pleural effusion, et al.
Long-term outcome | 5 years
  Total survival time after proximal gastrectomy for gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China